CLINICAL TRIAL: NCT06064474
Title: Effects of High Ventilation Breathwork With Retention (HVBR) on Mental Health and Wellbeing: A Randomised Placebo-controlled Trial
Brief Title: Effects of High Ventilation Breathwork With Retention (HVBR) on Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Collaborators: Sylff Association (Unknown); Brighton & Sussex Medical School (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Guy Fincham, Principal Investigator, University of Sussex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sussex fast breathwork study
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Stress; Anxiety; Depressive Symptoms; Mental Wellbeing; Positive Affect; Negative Affect; Sleep-Related Impairment
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High ventilation breathwork with retention (HVBR) (Experimental): Guided audio of HVBR pre-recorded by a trained breathwork facilitator for ~20min/day over 21 days (three weeks). Delivered remotely through audio link, comprising evocative music and four rounds of hyperventilation with four separate retentions (breath holds), progressively increasing in length (from ~45seconds up to ~90 seconds).
  Interventions: Behavioral: High ventilation breathwork with retention (HVBR)
- Placebo HVBR (Placebo Comparator): Guided audio of placebo HVBR pre-recorded by a trained breathwork facilitator for ~20min/day over 21 days (three weeks). Delivered remotely through audio link, comprising music and four rounds of paced breathing at 15b/min (equal inhale:exhale) with four separate brief retentions, progressively increasing in length (from ~10secs to ~25secs).
  Interventions: Behavioral: Placebo HVBR

INTERVENTIONS:
Behavioral: High ventilation breathwork with retention (HVBR) — Intervention
  Arms: High ventilation breathwork with retention (HVBR)
Behavioral: Placebo HVBR — Placebo
  Arms: Placebo HVBR

SUMMARY:
The investigators are conducting a randomised-controlled trial comparing high ventilation breathwork with retention (HVBR) to a breathwork placebo (paced breathing at 15breaths/min with brief retentions). The metric of 15b/min aligns with guidance from the British Journal of Nursing, Royal College of Physicians and Johns Hopkins Medicine which state that the average, healthy rate should range from: 12-20, 12-18 and 12-16b/min, respectively. The main questions the study attempts to address are: Does HVBR lead to improved state and trait mental health and wellbeing in a general population adult sample?

The study will be conducted entirely online through the research platform Prolific, so participant data will be anonymous. The investigators will collect self-reports of mental health and wellbeing before and after the three-week breathwork period, in addition to a follow-up three weeks later. Pre-post intervention and follow-up questionnaires will be completed online via the survey platform Qualtrics which will be linked to Prolific. Data on self-reported adherence to, and credibility/expectancy of, the breathwork will also be collected, along with participants' experiences to gauge the safety and tolerability of the breathwork protocol.

ELIGIBILITY:
Inclusion Criteria (self-assessed):

* Fluent in English and living in the UK
* Have access to headphones
* Comfortable with faster breathing and holding breath
* Willing to only practice breathwork in safe environment, lying down in soft area (i.e., bed, sofa, carpet/mat), and always away from water & hard ground
* Willing to only practice the breathwork away from large meals (i.e., before or 1hour after) and bedtime (i.e., at least 1 hour before if practicing in evening)

Exclusion Criteria (self-assessed):

* Hypotension or hypertension (low or high blood pressure)
* History of respiratory or cardiovascular/heart problems or disease
* History of fainting or syncope
* Epilepsy or seizures
* History of panic disorder or panic attacks
* Cerebral aneurysm
* Have had problems with prior breathwork sessions (i.e., fainting)
* Pregnancy, think one might be pregnant, trying to get pregnant, or are breastfeeding
* Any problems which affect one's ability to pace their breathing (i.e., active/chronic respiratory infection including blocked nose/cough/cold/fever, etc.), breathlessness, abnormally slow breathing (bradypnea), or abnormally fast breathing (tachypnoea)
* Any other physical/mental health conditions or current life events which impair or affect one's ability to engage in activities involving breath control
* Are taking any regular medication other than the contraceptive pill, including medications to reduce blood pressure (i.e., Ramipril or other ACE-inhibitors), beta blockers (i.e., Propranolol), antidepressants, anxiolytics or any other psychotropic medications

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Subjective stress | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and three weeks after the intervention). Primary timepoint is post-intervention
  Depression Anxiety Stress Scale-21 (DASS-21) - stress subscale (score range: 0-21; higher scores denote worse outcome). Score on DASS-21 then multiplied by two to convert it to the longer form DASS-42 final score

SECONDARY OUTCOMES:
Subjective anxiety | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and three weeks after the intervention)
  DASS-21 - anxiety subscale (score range: 0-21; higher scores denote worse outcome)
Subjective depressive symptoms | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and three weeks after the intervention)
  DASS-21 - depression subscale (score range: 0-21; higher scores denote worse outcome)
Subjective mental wellbeing | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and three weeks after the intervention)
  Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) (score range: 7 to 35; higher scores denote better outcome). Total raw scores are then transformed into metric scores using the SWEMWBS conversion table on: www.warwick.ac.uk
Subjective sleep-related impairment | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and three weeks after the intervention)
  PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 4a (score range: 5-20; higher scores denote worse outcome). Data scored using a T-score transformation according to PROMIS Sleep scoring manual on: www.healthmeasures.net
Subjective positive affect | Pre-intervention (immediately before the intervention), post first breathwork session (immediately after starting breathwork), and post-intervention (immediately after the intervention)
  Positive and Negative Affect Schedule (PANAS) positive affect subscale (score range: 10-50; higher scores denote better outcome)
Subjective negative affect | Pre-intervention (immediately before the intervention), post first breathwork session (immediately after starting breathwork), and post-intervention (immediately after the intervention)
  PANAS negative affect subscale (score range: 10-50; higher scores denote worse outcome)
Subjective credibility and expectancy of protocol | Immediately after starting breathwork intervention
  Credibility/Expectancy Questionnaire (CEQ-6). Two Sets (Credibility of course/therapy [breathwork] and expectancy of course/therapy [breathwork]). Four items scored 1-9 and two items scored 0-100%. Scores for expectancy set then standardised via converting them to z-scores. Higher scores denote greater credibility and/or expectancy of specific breathwork technique
Negative side effects due to protocol | Post-intervention (immediately after the intervention)
  Whether participants experienced unpleasant/unwanted short-term effects and/or lasting bad effects from the breathwork
Self-reported adherence to protocol | Post-intervention (immediately after the intervention)
  Number of sessions participants self-report practicing out of 21 days assigned

OTHER OUTCOMES:
Overall experience | Post-intervention and follow-up (immediately after the intervention, and three weeks after the intervention)
  Participants' perspectives and overall experience of the protocol/study-period
Hypothesis guessing | Follow-up (three weeks after the intervention)
  Whether participants can correctly guess which condition they were allocated to

CONTACTS AND LOCATIONS:
Overall Officials: Guy W Fincham, MSc, Principal Investigator — University of Sussex
Locations (1):
- Prolific, Remote/Online, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All participant data will be anonymous (only Prolific user IDs will be seen). No identifiable personal information will be collected. Participants will be able to check a box if they are happy for our research team at the University of Sussex to include the data again in future studies related to breathwork and meditation, as well as share with other research groups, if these have gained independent ethical approval, based on the strict confidentiality terms described in the participant info/consent form.
Supporting Information: Study Protocol, SAP
Time Frame: Indefinitely after the study has been completed.
Access Criteria: Our research team at the University of Sussex will have access. The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request to other researchers working on breathwork and meditation.

DOCUMENTS (2):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT06064474/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT06064474/SAP_001.pdf